CLINICAL TRIAL: NCT06583382
Title: Risk for Second Revision in Patients With Cemented Versus Non-cemented Acetabular Component at Primary THA. A National Cohort Study From DHR
Brief Title: Cementation of Cup and the Risk of Second Revision
Status: Not yet recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Saber Muthanna Saber, Principal Invistigator, Bispebjerg Hospital
Other Study IDs: P-2022-717
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Total Hip Arthroplasty (THA); Revision Hip Arthroplasty
Keywords: Cup cementation; total hip arthroplasty; THA; Revision; Second Revision; Re-revision; cement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cemented Cup: Patients who received a cemented acetabular component in their primary THA and underwent a revision surgery of the component
- Uncemented Cup: Patients who received an uncemented acetabular component in their primary THA and underwent a revision surgery of the component

SUMMARY:
Background:

The fixation method of the acetabular component during the primary total hip arthroplasty (THA) affects the surgical techniques implemented in the revision surgery and may influence the risk of second revision.

Objectives:

The objectives of this study are to investigate the risk of second revision of the cup alone or any component after first cup revision following cemented or non-cemented cup in the primary THA.

Methods/design:

The study is a nationwide register-based cohort study and will follow the reporting of studies Conducted using Observational Routinely collected health Data (RECORD) guidelines. We will compare the risk of undergoing a second revision between cemented and uncemented revised acetabular component by reporting the absolute risk of second revision of 1) the acetabular component and 2) any other component. The cumulative incidence of revision will be estimated using Fine-Gray regression to model the cumulative incidence function, accounting for the competing risk of death. We will apply both a crude and a multivariable adjusted model adjusting for age, sex, Charlson Comorbidity Index (CCI) and the 5-year intervals during which the primary operation was performed.

DETAILED DESCRIPTION:
Background Total hip arthroplasty (THA) is considered to be one of the most successful operations performed in orthopedic surgery and the treatment of choice for end-stage osteoarthritis of the hip. The frequency of revision surgery for total hip joint arthroplasty continues to increase worldwide. Generally, the longevity of revision THA is less than that of primary THA. Although the optimal component fixation method in primary THA is still debated, several studies have shown increased use of the cementless technique in most parts of the world. The use of cementless technology in THA initially gained popularity as complications such as aseptic loosening and "cement disease" began to surface with the use of first-generation cement techniques. Cementless acetabular components have achieved widespread acceptance in THA as a result of their improved and reliable long-term results. Primary stability is achieved through press-fit fixation that requires 1-3 mm under-reaming of the acetabular cavity and forceful impaction. Studies have shown slightly higher risk of revision in uncemented acetabular components compared to those cemented. We believe that the differences in the fixation method during the primary operation significantly affects the surgical techniques implemented in the first revision of each group and by that influencing the risk of second revision. This was shown before in cemented vs. uncemented stem, but no study has to our knowledge reported the same concerning acetabular components. In previous studies comparing the risk of revision in patients undergoing THA with cemented and hybrid fixation techniques (where the cup component is non-cemented), the hybrid technique was associated with a higher risk of revision for any reason compared to the cemented technique, regardless of the patient's sex and age. The justification for this difference in revision rates can be the use of cement in cup fixation. This suggests that the use of cement in cup fixation may provide certain advantages, such as increased stability or longevity, which could potentially lead to a lower risk of revision compared to non-cemented cup fixation. Therefore, further research and clinical considerations are necessary to fully understand the implications of cup fixation techniques in risk of THA revision. We expect that the result from this study would help in the choice of fixation technique by shedding light on an under investigated outcome concerning the complications associated with fixation technique.

Objective The objectives of this study are to investigate the risk of second revision of the cup alone or any component after first cup revision following cemented or non-cemented cup in the primary THA.

Methods Study design The current study is a nationwide register-based cohort study that utilizes prospectively collected data from the Danish Hip Arthroplasty Register (DHR) and the Danish National Patient Registry (DNPR). The study will follow the reporting of studies Conducted using Observational Routinely collected health Data (RECORD) guidelines. We will include patients who have undergone THA at both public and private hospitals from January, 1st ,1995, to December 31st, 2020, to ensure a minimum follow-up of 1 year. Patients will be followed from the date of the first revision and until the first of the following: Implant removal of the acetabular component, death, emigration, until the date where there is a minimum of 100 patients left in the risk set for each group, or until December 31st, 2021.

Data sources and linkage We will use data from the DHR and the DNPR. The DHR was founded in 1995 prospectively collects data on all THAs in public and private hospitals and their subsequent revisions in Denmark. Reporting from both public and private hospitals is mandatory. As of 2021, the DHR has a reporting rate of 97% for primary THAs and 95% for revisions. The DNPR is a national administrative database that registers all hospital contacts, including discharge diagnoses. All Danish residents have a unique 10-digit Civil Personal Register (CPR) number in the Danish Civil Registration System (DCRS) and this number enables to cross-link inhabitants in Denmark across different databases and to be traced until death or emigration.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis as the indication for the primary THA.
* Has experienced a first revision with exchange of the liner, femoral head and/or acetabular component either with or without exchange of the femoral component.
* Femoral with a size of 28mm, 32mm or 36mm after the first revision
* Surgery with the posterior approach.

Exclusion Criteria:

* Isolated revision of the femoral component.
* Constrained liner.
* Metal-on-metal implant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include patients who have undergone THA at both public and private hospitals from January, 1st ,1995, to December 31st, 2020, to ensure a minimum follow-up of 1 year. Patients will be followed from the date of the first revision and until the first of the following: Implant removal of the acetabular component, death, emigration, until the date where there is a minimum of 100 patients left in the risk set for each group, or until December 31st, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The absolute risk of second revision of the cup | minimum of 1 year and a maximum of 15 years
  The absolute risk of undergoing a second revision of the acetabular component after having first revision with exchange of the acetabular component.
  Revision is defined as any surgical procedure that involves skin incision in the ipsilateral hip joint due to acetabular component failure as reported in the Danish hip register or having one of the following NOMESCO (Nordic Medico-Statistical Committee) Classification of Surgical Procedures codes in the DNPR: KNFC2, KNFC01, KNFC3, KNFC4, KNFC10, KNFC11,KNFC21, KNFC31, KNFC41, KNFC29, KNFC20, KNFC40, KNFC49

SECONDARY OUTCOMES:
The absolute risk of second revision of any other component | minimum of 1 year and a maximum of 15 years
  The absolute risk of undergoing a second revision of any other component after having first revision with exchange of the acetabular component. Revision is defined as any surgical procedure that involves skin incision in the ipsilateral hip joint due to acetabular component failure as reported in the Danish hip register or having one of the following NOMESCO (Nordic Medico-Statistical Committee) Classification of Surgical Procedures codes in the Danish national patient register: KNFC02, KNFC20, KNFC22, KNFC23, KNFC32, KNFC33, NFC42, KNFC43, KNFC59, KNFC99, KNFA0, KNFA1, KNFA2, KNFG09, KNFS19, KNFS49, NFS99, KNFW49, KNFW69, KNFW89, KNFW99, KNFW59, KNFW79, NFU1Y, NFU89, NFU99, NFT99, NFP29

CONTACTS AND LOCATIONS:
Overall Officials: Søren Overgard, MD, PhD, DMSc, Study Director — Department of Orthopedic surgery and traumatology, Hvidovre Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT06583382/Prot_SAP_000.pdf